CLINICAL TRIAL: NCT04385381
Title: A Clinical Study Investigating the Safety and Efficacy of the URECA CTO Device
Brief Title: Safety and Efficacy of the URECA CTO Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: change of manufacterer of medical device
Sponsor: Ureca BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URECA
Record Dates: First submitted 2020-05-06; First posted 2020-05-12 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Intervention Model Description: facilitating guidewire re-entry into the true lumen after passing occlusion(s) in the peripheral vasculature with the URECA CTO device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- URECA CTO device (Experimental): investigate the safety and efficacy of the URECA CTO device in facilitating guidewire re-entry into the true lumen after passing occlusion(s) in the peripheral vasculature.
  Interventions: Device: URECA CTO device

INTERVENTIONS:
Device: URECA CTO device — facilitating guidewire re-entry into the true lumen after passing occlusion(s) in the peripheral vasculature with the URECA CTO device.

SUMMARY:
Clinical study to investigate the safety and the efficacy of the URECA CTO Device during recanalization and mechanical re-entry into the true lumen after passing the occlusions/calcifications (chronic total occlusions) in the peripheral vasculature.

DETAILED DESCRIPTION:
Peripheral Arterial Disease (PAD) restricts blood supply to the lower limbs. The disease causes obstructions that can affect blood vessels in both the proximal and distal regions. When these vessel obstructions exist for more than 3- 6 Months they are classed as chronic total occlusions. Without sufficient collateral formation this can lead to to chronic limb-treatening ischemia (CLTI), which is characterized by chronic pain and tissue loss. Without revascularization this frequently leads to amputation. The purpose of this clinical study is to investigate the safety and the efficacy of the URECA CTO Device during recanalization and mechanical re-entry into the true lumen after passing the occlusions/calcifications (chronic total occlusions) in the peripheral vasculature.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be >= 18 and <= 85 years old
* Clinically diagnosed for endovascular treatment of peripheral vascular disease and chronic total occlusion in the iliac artery, superficial femoral artery or in the proximal popliteal artery determined by duplex, CTA, MRA and/or DSA.
* Patient has been assessed by an independent vascular surgeon and an interventional radiologist.
* Written and signed informed consent

Exclusion Criteria:

* 1. Concomitant hepatic insufficiency, thrombophlebitis, deep venous thrombus, coagulation disorder or receiving immunosuppressant therapy; 2. Severe infection or soft tissue loss that may preclude any meaningful attempt at limb salvage; 3. Known or suspected allergies or contraindications to contrast agents; 4. Any significant medical condition which, in the investigator's opinion, may interfere with the subject's optimal participation in the study; 5. The subject is currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study; 6. Patient unable to give consent; 7. Pregnant and breastfeeding women; 8. Patients who recently suffered from a stroke and/or a myocardial infarct (Within 2 months) 9. Patients with an uncontrollable diabetes; 10. Severe intercurrent illness that, in the opinion of the investigator, may put the subject at risk when participating in the study 11. Patients with hypercoagulopathy; 12. Stent in place in the to be treated artery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
device success, | during surgery
  the successful placement of a guidewire in the true lumen distal of the CTO using the URECA CTO Device without the occurrence of device related complications that involve a Serious Adverse Event.
safety of device | 6 weeks after surgery
  absence of device related Serious Adverse Events.

SECONDARY OUTCOMES:
Adverse Events | 6 weeks after surgery
  device related complications that involve a Adverse Event.
procedure time | during surgery
  time whole procedure takes using the URECA CTO device
Total Fluoroscopy Time and | during surgery
  The amount of time of fluoroscopy between the time of introducer sheath puncture up to the moment of sheath removal
Total Contrast Load | during surgery
  the amount of contrast load between the time of introducer sheath puncture up to the moment of sheath removal

CONTACTS AND LOCATIONS:
Overall Officials: JW Kuiper, MD, Principal Investigator — Ikazia Ziekenhuis
Locations (1):
- Ikazia ziekenhuis, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No